CLINICAL TRIAL: NCT01642784
Title: Complete Infarct Related Artery Revascularization in Acute Myocardial Infarction Registry(CORAMIreg)
Brief Title: Complete Infarct Related Artery Revascularization in Acute Myocardial Infarction
Acronym: CORAMIreg
Status: Completed | Type: Observational
Sponsor: Fundacja Ośrodek Badań Medycznych (Other)
Responsible Party: Sponsor
Other Study IDs: 2.0, 2011-11-24
Record Dates: First submitted 2012-06-25; First posted 2012-07-17 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Myocardial Infarction
Keywords: STEMI; NSTEMI; revascularization; stents
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Culprit lesion IRA revascularization: Culprit lesion IRA revascularization
  Interventions: Device: Primary PCI of culprit lesion in IRA with drug eluting stent (DES)
- Complete IRA revascularization: Complete IRA revascularization
  Interventions: Device: Primary PCI of culprit lesion in IRA with drug eluting stent (DES) and PCI of the other critical lesion in IRA with another DES

INTERVENTIONS:
Device: Primary PCI of culprit lesion in IRA with drug eluting stent (DES) — Primary PCI of culprit lesion in IRA with drug eluting stent (DES)
  Groups: Culprit lesion IRA revascularization
Device: Primary PCI of culprit lesion in IRA with drug eluting stent (DES) and PCI of the other critical lesion in IRA with another DES — Primary PCI of culprit lesion in IRA with drug eluting stent (DES) and PCI of the other critical lesion in IRA with another DES
  Groups: Complete IRA revascularization

SUMMARY:
Objective of this registry study is to compare strategy of complete vs. target lesion-only primary PCI (percutaneous coronary intervention) in IRA (infarct related artery) in STEMI (ST elevation myocardial infarction) patients.

DETAILED DESCRIPTION:
CORAMI is a registry study addressing the issue of complete vs culprit-only PCI within infarct related artery in patients with ST-elevation and non-ST elevation myocardial infarction treated with interventional procedures.

The main objectives of the study include:

1. gathering data on patients with at least two independent critical stenotic lesions in IRA (one of which is the culprit lesion) during index primary PCI for STEMI or NSTEMI (prevalence, characteristic, predisposing factors).
2. comparing chosen treatment strategies for multiple lesion IRA
3. comparison of complete vs. target lesion-only PCI in IRA in acute MI (myocardial infarction) patients.

The study clinical hypothesis is that stenting single critical - culprit lesion in multi-lesion IRA in MI patients during index PCI procedure is superior to stenting all critical lesions in IRA in terms of early treatment result and might be associated with less frequent periprocedural angiographic complications.

H0: The efficacy in terms of early treatment result of stenting one critical - culprit lesion in multilesions IRA in acute MI patients is less or equal to efficacy of stenting all critical lesions in IRA.

H1: The efficacy in terms of early treatment result of stenting one critical - culprit lesion in multilesions IRA in acute MI patients is greater than efficacy of stenting all critical lesions in IRA.

CORAMI Registry is a prospective, international (Poland, Slovenia), multicenter observational study with retrospective chart review which will be performed in experienced invasive facility centres with 24/7 PCI duty and continuous patient enrollment for 18 months (January 2011 - June 2012).

This study will collect data on all consecutive patients with STEMI and NSTEMI undergoing immediate coronary angiography which demonstrated at least two independent (requiring two stent platforms) critical lesions in infarct related artery (one of which is considered as target/culprit lesion that have caused the myocardial infarction and requires immediate PCI). Patients will be treated (multiple or single lesion stenting) according to local standard and operator's decision. Patient follow up phone call and/or visit (according to local protocols) will be performed at 12 months from enrollment if applicable by local standards.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of STEMI or NSTEMI (according to ESC 2007 definition)
* Over 18 years of age
* Presence of two critical lesions requiring PCI in IRA (LAD (left anterior descending), Cx (circumflex), RCA (right coronary artery)):

  1. Target/culprit lesion which requires immediate stenting (>50 - 100%) and
  2. Second critical lesion (70-90%).

Exclusion Criteria:

* Terminal illness with life expectancy less <1 year or active cancer disease,
* Pregnancy or possibility of pregnancy
* Second critical lesion in IRA >90% or occlusion
* Contraindications to PCI or/and stent implantation
* Con-current participation in another clinical study that did not meet its primary end-point

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will comprise of approx. 200 patients (males and females) with the diagnosis of STEMI or NSTEMI and at least two independent critical lesions in infarct related artery (one of which is considered as target/culprit lesion that have caused the myocardial infarction and requires immediate PCI). Patients enrolled to the registry must meet all the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Death | At 12 months
  Death rates at 12-month clinical follow-up
Stent thrombosis | At 12 months
  Rates of stent thrombosis at 12-month follow-up according to ARC definition
reMI (repeat myocardial infarctions) | At 12 months
  Rates of reMI at 12 months
urgent TVR (target vessel revascularization) at 12 months | 12 months and at 12 months
  Rates of urgent TVR at 12 months
Planned TVR | At 12 months
  Rates of planned TVR (PCI + CABG) at 12 months

SECONDARY OUTCOMES:
Angiographic complications | During hospitalization
  Immediate in-hospital angiographic complications (at least one or more of the following: distal embolisation, no-reflow, slow-flow, acute coronary artery occlusion, artery perforation, tamponade, dissection type B and above)
Target Vessel Revascularization (PCI and/or CABG (coronary artery bypass graft)) | During hospitalization and at 12 months
  Urgent in-hospital Target Vessel Revascularization (PCI and/or CABG)
Complete contrast dose in ml | During hospitalization and at 12 months
  Complete contrast dose in ml
Complete radiation dose in mGy | During hospitalization and at 12 months
  Complete radiation dose in mGy

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Januś, MD, PhD, Principal Investigator — Pracownia Hemodynamiki Szpital im. E. Szczeklika
Locations (8):
- Poland (7):
  - Krakowskie centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Carint Scanmed Sp. z o.o., Krakow
  - Centrum Kardiologii Inwazyjnej GVM Carint, Ostrowiec Świętokrzyski
  - Centrum Kardiologii Inwazyjnej GVM Carint, Oświecim
  - Oddział Kardiologii Inwazyjnej, Elektroterapii i Angiologii w Pińczowie, Pińczów
  - Podkarpackie Centrum Interwencji Sercowo -Naczyniowych NZOZ, Sanok
  - Pracownia Hemodynamiki Szpital im. E. Szczeklika, Tarnów
  - I Katedra i Klinika Kardiologii, Warszawski Uniwersytet Medyczny, Warsaw
- Departament of Cardiology, University Hospital, Ljubljana, Ljubljana, Slovenia